CLINICAL TRIAL: NCT02869789
Title: A Phase 3b/4 Safety Trial of Flat Dose Nivolumab In Combination With Ipilimumab in Participants With Non-Small Cell Lung Cancer
Brief Title: An Investigational Immuno-therapy Study for Safety of Nivolumab in Combination With Ipilimumab to Treat Advanced Cancers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-817; 2016-002621-10 (EudraCT Number)
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab in combination with Ipilimumab (Experimental): Specified dose on specified days
  Interventions: Drug: Nivolumab in combination with Ipilimumab

INTERVENTIONS:
Drug: Nivolumab in combination with Ipilimumab — Specified dose on specified days
  Other Names: BMS-936558 (Nivolumab); Opdivo (Nivolumab); BMS-734016 (Ipilimumab); Yervoy (Ipilimumab)

SUMMARY:
A study to evaluate the safety of Nivolumab given in combination with Ipilimumab in patients with advanced cancers. The initial group will enroll patients with newly diagnosed Stage 4 or non-small cell lung cancer that has come back.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage 4 or recurrent non-small cell lung cancer
* Eastern Cooperative Oncology Group (ECOG) score 0-1 (Physically able to carry out light housework or office work through to being fully active as you were before cancer)
* No prior systemic anticancer therapy (including EGFR and ALK inhibitors)
* Tissue or Programmed death-ligand 1 (PD-L1) results available

Cohort 1A Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) score 2 or
* Eastern Cooperative Oncology Group (ECOG) score 0-1 and one disease specific criteria as listed in the protocol

Cohort C Inclusion Criteria:

* High Tumor Mutation Burden

Exclusion Criteria:

* Untreated brain metastases
* An active malignancy that requires concurrent intervention
* Active, known or suspected autoimmune disease
* Carcinomatous meningitis, which means there is inflammation of the covering of the brain, caused by cancer

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1041 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (136):
- United States (61):
  - Local Institution - 0121, Birmingham, Alabama
  - Local Institution - 0148, Phoenix, Arizona
  - Local Institution - 0085, Tucson, Arizona
  - Local Institution - 0164, Little Rock, Arkansas
  - Local Institution - 0146, Bakersfield, California
  - Marin Cancer Care, Inc, Greenbrae, California
  - Los Angeles Hematology/Oncology Medical Group, Los Angeles, California
  - Local Institution - 0115, Los Angeles, California
  - Torrance Health Association, Redondo Beach, California
  - Va San Diego Healthcare System, San Diego, California
  - Local Institution - 0143, San Luis Obispo, California
  - Local Institution - 0144, Santa Maria, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Local Institution - 0161, Whittier, California
  - Local Institution - 0083, Denver, Colorado
  - Local Institution - 0141, Grand Junction, Colorado
  - Cancer Specialists of North FL, Jacksonville, Florida
  - Local Institution - 0082, Ocala, Florida
  - Local Institution - 0147, Pembroke Pines, Florida
  - Local Institution - 0163, Athens, Georgia
  - Local Institution - 0002, Atlanta, Georgia
  - Local Institution - 0166, Atlanta, Georgia
  - Local Institution - 0088, Niles, Illinois
  - Local Institution - 0108, Wichita, Kansas
  - Kentucky One Health St. Joseph East Cancer Center, Lexington, Kentucky
  - Local Institution - 0091, Columbia, Maryland
  - Local Institution - 0089, Edina, Minnesota
  - Jackson Oncology Associates, Pllc, Jackson, Mississippi
  - Local Institution - 0077, Grand Island, Nebraska
  - Local Institution - 0087, Las Vegas, Nevada
  - Local Institution - 0170, Reno, Nevada
  - Local Institution - 0156, Belleville, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Local Institution - 0142, Livingston, New Jersey
  - Local Institution - 0167, The Bronx, New York
  - Local Institution - 0004, Durham, North Carolina
  - Local Institution - 0012, Winston-Salem, North Carolina
  - Local Institution - 0100, Cincinnati, Ohio
  - Local Institution - 0134, Cleveland, Ohio
  - Local Institution - 0172, Corvallis, Oregon
  - Local Institution - 0096, Eugene, Oregon
  - Local Institution - 0176, Portland, Oregon
  - Local Institution - 0139, Allentown, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Local Institution - 0159, Pittsburgh, Pennsylvania
  - Local Institution - 0001, Sayre, Pennsylvania
  - Local Institution - 0123, Charleston, South Carolina
  - Local Institution - 0066, Chattanooga, Tennessee
  - Local Institution - 0067, Nashville, Tennessee
  - Local Institution - 0090, Austin, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Local Institution - 0149, Dallas, Texas
  - Local Institution - 0094, Fort Worth, Texas
  - Local Institution - 0093, Longview, Texas
  - Local Institution - 0098, Plano, Texas
  - Local Institution - 0086, Waco, Texas
  - Local Institution - 0097, Fairfax, Virginia
  - Local Institution - 0044, Richmond, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Local Institution - 0174, Renton, Washington
  - Local Institution - 0173, Spokane, Washington
- Argentina (5):
  - Local Institution - 0008, Capital Federal, Buenos Aires
  - Local Institution - 0006, Viedma, Río Negro Province
  - Local Institution - 0007, CABA
  - Local Institution - 0009, Córdoba
  - Local Institution - 0126, San Miguel de Tucumán
- Belgium (3):
  - Local Institution - 0038, Ghent
  - Local Institution - 0037, Liège
  - Local Institution - 0036, Sint-Niklaas
- Brazil (4):
  - Local Institution - 0152, Ijuí, Rio Grande do Sul
  - Local Institution - 0154, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0153, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0151, Barretos, São Paulo
- Canada (4):
  - Local Institution - 0127, Greenfield Park, Quebec
  - Local Institution - 0109, Montreal, Quebec
  - Local Institution - 0049, Rimouski, Quebec
  - Local Institution - 0050, Trois-Rivières, Quebec
- Chile (2):
  - Local Institution - 0010, Santiago, Santiago Metropolitan
  - Local Institution - 0011, Santiago
- Czechia (2):
  - Local Institution - 0133, Nový Jičín
  - Local Institution - 0130, Prague
- France (9):
  - Local Institution - 0118, Bordeaux
  - Local Institution - 0075, Dijon
  - Local Institution - 0069, Marseille
  - Local Institution - 0076, Paris
  - Local Institution - 0074, Pessac
  - Local Institution - 0071, Rennes
  - Local Institution - 0070, Saint-Herblain
  - Local Institution - 0072, Strasbourg
  - Local Institution - 0073, Toulon
- Germany (5):
  - Local Institution - 0023, Frankfurt
  - Local Institution - 0028, Gera
  - Local Institution - 0029, Kassel
  - Local Institution - 0026, Löwenstein
  - Local Institution - 0025, Wiesbaden
- Greece (3):
  - Local Institution - 0030, Athens
  - Local Institution - 0031, N. Faliro
  - Local Institution - 0032, Thessaloniki
- Hungary (2):
  - Local Institution - 0013, Gyöngyös - Mátraháza, Heves County
  - Local Institution - 0014, Budapest
- Italy (8):
  - Local Institution - 0054, Milan, Lombardy
  - Ospedale Policlinico San Martino, Genova
  - IRST Meldola, Meldola
  - AOU della Campania Luigi Vanvitelli, Napoli
  - Local Institution, Napoli
  - Ospedale Degli Infermi, Rimini
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda Ospedaliera Santa Maria Terni, Terni
- Local Institution - 0019, Monterrey, NL, Mexico
- Netherlands (2):
  - Local Institution - 0045, Groningen
  - Local Institution - 0035, Rotterdam
- Poland (3):
  - Local Institution - 0015, Bydgoszcz
  - Local Institution - 0068, Sucha Beskidzka
  - Local Institution - 0016, Warsaw
- Romania (3):
  - Local Institution - 0128, Bucharest
  - Local Institution - 0119, Craiova
  - Local Institution - 0120, Romania
- Russia (3):
  - Local Institution - 0022, Moscow
  - Local Institution - 0021, Moscow
  - Local Institution - 0020, Saint Petersburg
- Spain (8):
  - Local Institution - 0061, A Coruña
  - Local Institution - 0060, Barcelona
  - Local Institution - 0062, Jaén
  - Local Institution - 0065, Madrid
  - Local Institution - 0064, Majadahonda - Madrid
  - Local Institution - 0063, Seville
  - Local Institution - 0059, Valencia
  - Local Institution - 0112, Zaragoza
- Switzerland (2):
  - Local Institution - 0048, Basel
  - Local Institution - 0046, Zurich
- Local Institution - 0104, Antalya, Turkey (Türkiye)
- United Kingdom (5):
  - Local Institution - 0041, London, Greater London
  - Local Institution - 0039, Leicester, Leicestershire
  - Local Institution - 0040, Edinburgh, Midlothian
  - Local Institution - 0042, Metropolitan Borough of Wirral
  - Local Institution - 0043, Newcastle upon Tyne

REFERENCES:
- [Derived] Ready NE, Audigier-Valette C, Goldman JW, Felip E, Ciuleanu TE, Rosario Garcia Campelo M, Jao K, Barlesi F, Bordenave S, Rijavec E, Urban L, Aucoin JS, Zannori C, Vermaelen K, Aren Frontera O, Curioni Fontecedro A, Sanchez-Gastaldo A, Juan-Vidal O, Linardou H, Poddubskaya E, Spigel DR, Ahmed S, Maio M, Li S, Chang H, Fiore J, Acevedo A, Paz-Ares L. First-line nivolumab plus ipilimumab for metastatic non-small cell lung cancer, including patients with ECOG performance status 2 and other special populations: CheckMate 817. J Immunother Cancer. 2023 Feb;11(2):e006127. doi: 10.1136/jitc-2022-006127. PMID 36725084
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Analysis for the NSCLC special population cohort A1 is pre-specified as exploratory.
Groups:
- Cohort A: First-line NSCLC: Nivolumab 240 mg IV Q2W + Ipilimumab 1 mg/kg IV Q6W, starting on Day 1, until progression, unacceptable toxicity, withdrawal of consent, 24 months of treatment from the first dose, or the study ends, whichever occurs first
- Cohort A1: First-line NSCLC special population: Nivolumab 240 mg IV Q2W + Ipilimumab 1 mg/kg IV Q6W, starting on Day 1, until progression, unacceptable toxicity, withdrawal of consent, 24 months of treatment from the first dose, or the study ends, whichever occurs first
- Cohort B: Second-line NSCLC: Nivolumab 240 mg IV Q2W + Ipilimumab 1 mg/kg IV Q6W, starting on Day 1, until progression, unacceptable toxicity, withdrawal of consent, 24 months of treatment from the first dose, or the study ends, whichever occurs first
- Cohort C: First-line NSCLC high tumor mutational burden (H-TMB >= 10 mutations/MB): Nivolumab 240 mg IV Q2W + Ipilimumab 1 mg/kg IV Q6W, starting on Day 1, until progression, unacceptable toxicity, withdrawal of consent, 24 months of treatment from the first dose, or the study ends, whichever occurs first
Period: Overall Study
Arm/Group | Cohort A | Cohort A1 | Cohort B | Cohort C
Started | 391 | 198 | 395 | 57
Completed | 56 | 16 | 30 | 12
Not Completed | 335 | 182 | 365 | 45
Not completed — Disease progression | 184 | 109 | 260 | 19
Not completed — Study drug toxicity | 90 | 32 | 55 | 14
Not completed — Death | 7 | 3 | 5 | 1
Not completed — Adverse Event unrelated to study drug | 30 | 18 | 21 | 6
Not completed — Participant request to discontinue study treatment | 10 | 5 | 5 | 3
Not completed — Withdrawal by Subject | 5 | 2 | 7 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Maximum clinical benefit | 5 | 2 | 1 | 0
Not completed — Poor/Non-compliance | 0 | 2 | 1 | 0
Not completed — Participant no longer meets study criteria | 0 | 1 | 1 | 0
Not completed — Administrative reason by sponsor | 0 | 0 | 1 | 0
Not completed — Other reasons | 4 | 8 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort A1 | Cohort B | Cohort C | Total
Number analyzed (Participants) | 391 | 198 | 395 | 57 | 1041
Age, Customized [Number; unit: Participants]
  < 65 years old | 183 | 81 | 200 | 24 | 488
  >= 65 and < 85 years old | 206 | 115 | 195 | 30 | 546
  >= 85 years old | 2 | 2 | 0 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 71 | 128 | 29 | 383
  Male | 236 | 127 | 267 | 28 | 658
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 13 | 12 | 3 | 38
  Not Hispanic or Latino | 185 | 78 | 175 | 54 | 492
  Unknown or Not Reported | 196 | 107 | 208 | 0 | 511
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 4 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 5 | 8 | 22
  White | 379 | 194 | 382 | 47 | 1002
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With High Grade (Grade 3-4 and Grade 5) Drug-Related Select Adverse Events (AEs)
Description: Drug related AEs are those events with relationship to study drug. If the relationship to study drug is missing, the AE will be considered as drug-related. The select AEs of interest are the following: Pulmonary, Renal, Gastrointestinal, Hepatic, Skin, Endocrine, and hypersensitivity/infusion reaction events. AEs are reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.
  Grade 3= Prolonged severe reaction Grade 4= Life threatening Grade 5= Death
Time Frame: From first dose to 30 days post last dose (Up to approximately 27 months)
Population: All treated participants as pre-specified in Cohort A, B, and C
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 391 | 395 | 57
Participants
  Gastrointestinal AEs grade 3-4 | 19 | 15 | 4
  Gastrointestinal AEs grade 5 | 0 | 0 | 0
  Hepatic AEs grade 3-4 | 25 | 17 | 3
  Hepatic AEs grade 5 | 0 | 0 | 0
  Pulmonary AEs grade 3-4 | 18 | 11 | 2
  Pulmonary AEs grade 5 | 0 | 1 | 0
  Renal AEs grade 3-4 | 2 | 1 | 1
  Renal AEs grade 5 | 0 | 0 | 0
  Skin AEs grade 3-4 | 14 | 9 | 2
  Skin AEs grade 5 | 0 | 0 | 0
  Endocrine AEs grade 3-4 | 16 | 11 | 2
  Endocrine AEs grade 5 | 0 | 0 | 0
  Hypersensitivity/Infusion Reaction grade 3-4 | 6 | 3 | 0
  Hypersensitivity/Infusion Reaction grade 5 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With High Grade (Grade 3-4 and Grade 5) Immune-Mediated Adverse Events (imAEs)
Description: imAEs are specific events that include pneumonitis, diarrhea/colitis, hepatitis, nephritis/renal dysfunction, rash, and endocrine (adrenal insufficiency, hypothyroidism/thyroiditis, hyperthyroidism, diabetes mellitus, and hypophysitis). AEs are reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.
  Grade 3= Prolonged severe reaction Grade 4= Life threatening Grade 5= Death
Time Frame: From first dose to 100 days post last dose (Up to approximately 29 months)
Population: All treated participants as pre-specified in Cohort A, B, and C
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 391 | 395 | 57
Participants
  Pneumonitis grade 3-4 | 20 | 14 | 3
  Diarrhea/Colitis grade 3-4 | 19 | 15 | 3
  Hepatitis grade 3-4 | 18 | 13 | 1
  Adrenal Insufficiency grade 3-4 | 5 | 4 | 1
  Hypothyroidism/Thyroiditis grade 3-4 | 2 | 2 | 0
  Hypothyroidism grade 3-4 | 1 | 1 | 0
  Thyroiditis grade 3-4 | 1 | 1 | 0
  Diabetes Mellitus grade 3-4 | 1 | 0 | 0
  Nephritis and Renal Dysfunction grade 3-4 | 2 | 1 | 0
  Rash grade 3-4 | 14 | 8 | 1
  Hypersensitivity grade 3-4 | 4 | 2 | 0
  Hyperthyroidism grade 3-4 | 0 | 2 | 0
  Hypophysitis grade 3-4 | 3 | 1 | 1
  Any category imAEs grade 5 | 0 | 0 | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from first dosing date to the date of the first documented tumor progression, as determined by investigators (per RECIST v1.1), or death due to any cause, whichever occurs first.
  Progressive Disease (PD)= ≥ 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an absolute increase of ≥ 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From first dosing date to the date of first documented tumor progression or, death due to any cause, whichever occurs first (Up to approximately 67 months)
Population: All treated participants as pre-specified in Cohort A, B, and C
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 391 | 395 | 57
Months | 5.75 [4.50 to 7.62] | 3.91 [2.89 to 4.24] | 11.10 [6.47 to 18.40]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first dosing date to the date of death. A participant who has not died will be censored at last known date alive.
Time Frame: From first dosing date to the date of death (Up to approximately 67 months)
Population: All treated participants as pre-specified in Cohort A, B, and C
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 391 | 395 | 57
Months | 16.76 [14.65 to 22.41] | 10.45 [8.84 to 12.22] | 26.09 [21.85 to NA] — Insufficient number of participants with events

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of confirmed complete response (CR) or partial response (PR).
  CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR= ≥ 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dosing date up to approximately 67 months
Population: All treated participants as pre-specified in Cohort A, B, and C
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 391 | 395 | 57
Percentage of participants | 37.3 [32.5 to 42.3] | 22.8 [18.7 to 27.2] | 45.6 [32.4 to 59.3]

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time between the date of first confirmed complete response (CR) or partial response (PR) to the date of the first documented tumor progression per RECIST 1.1, or death due to any cause, whichever occurs first.
  CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR= ≥ 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD)= ≥ 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an absolute increase of ≥ 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: as for outcome 3
Population: All treated participants with confirmed CR or PR as pre-specified in Cohort A, B, and C
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 146 | 90 | 26
Months | 27.56 [20.40 to 36.04] | 13.01 [10.12 to 19.29] | 26.05 [12.22 to NA] — Insufficient number of participants with events

7. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) Using Functional Assessment of Cancer Therapy-Lung (FACT-L)
Description: FACT-L is a quality-of-life questionnaire which includes Lung Cancer Subscale (LCS) that assesses the treatment impact on lung cancer related symptoms in 5 domains: Physical, social/family, emotional, and functional well-being using a 5-point scale (0=not at all; 1=a little bit, 2=somewhat; 3=quite a bit; 4=very much) added to obtain total score. The ranges of possible total scores are 0-136 for the FACT-L with a higher score representing better quality of life, improved symptomatology and enhanced physical/functional outcomes. According to Functional Assessment of Chronic Illness Therapy scoring guidelines, in the event of missing responses for some of the questions, scores will be prorated using the average of the other answers in that scale.
  Baseline is defined as events that occur before the date/time of first dose. Post treatment visits include follow-up (FU) visit 1, FU visit 2, and subsequent survival FU visits to occur every 3 months up until survival FU visit 18.
Time Frame: From baseline and up to subsequent survival follow-up visit 18 (Up to approximately 67 months)
Population: All treated participants who have an assessment at baseline and at least 1 follow-up assessment as pre-specified in Cohort A, B, and C
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 364 | 365 | 57
Units on a Scale
  Baseline | 94.89 (19.33) | 91.20 (18.45) | 93.96 (17.28)
  Treatment Week 6: number analyzed (Participants) | 245 | 244 | 41
  Treatment Week 6 | -0.84 (13.82) | -0.30 (14.87) | 2.72 (12.95)
  Survival Follow-up visit 6: number analyzed (Participants) | 22 | 16 | 2
  Survival Follow-up visit 6 | 14.68 (13.58) | 3.81 (18.59) | 12.42 (24.87)
  Survival Follow-up visit 16: number analyzed (Participants) | 3 | 1 | 0
  Survival Follow-up visit 16 | 5.28 (28.19) | -18.00 (NA) — Insufficient number of participants with events |
  Survival Follow-up visit 18: number analyzed (Participants) | 1 | 0 | 0
  Survival Follow-up visit 18 | -43.33 (NA) — Insufficient number of participants with events |  |

ADVERSE EVENTS:
Time Frame: SAEs and AEs are assessed from first dose to 100 days post last dose (Up to approximately 29 months). Participants were assessed for all-cause mortality from their first dose to their study completion (Up to approximately 67 months).
Arm/Group | Cohort A | Cohort A1 | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 294/391 | 166/198 | 334/395 | 32/57
Serious Adverse Events (participants affected / at risk) | 264/391 | 149/198 | 282/395 | 42/57
Other Adverse Events (participants affected / at risk) | 362/391 | 174/198 | 346/395 | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=391) | Cohort A1 (N=198) | Cohort B (N=395) | Cohort C (N=57)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4 | 2
Autoimmune anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 3 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 3 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 1 | 2 | 2
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 2 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 2
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 6 | 2 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 6 | 2 | 4 | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 2 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0
Euthyroid sick syndrome (Endocrine disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 3 | 0
Hypophysitis (Endocrine disorders) | 3 | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 1 | 0 | 1 | 0
Thyroiditis (Endocrine disorders) | 1 | 0 | 1 | 0
Ophthalmoplegia (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 5 | 3 | 6 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 11 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 3 | 4 | 5 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 2 | 1
Asthenia (General disorders) | 4 | 1 | 2 | 1
Chest pain (General disorders) | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 2 | 0 | 2 | 0
Disease progression (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 3 | 3 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 2 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 4 | 0
Performance status decreased (General disorders) | 1 | 1 | 3 | 0
Pyrexia (General disorders) | 5 | 8 | 7 | 0
Sudden death (General disorders) | 6 | 4 | 4 | 2
Ulcer (General disorders) | 0 | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 1 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 2 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 4 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 3 | 7 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Colonic abscess (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 4 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Fungal oesophagitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 1 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0
Infective spondylitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 21 | 6 | 26 | 2
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 7 | 4 | 3 | 0
Sepsis (Infections and infestations) | 7 | 4 | 5 | 2
Septic shock (Infections and infestations) | 5 | 2 | 2 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Incision site impaired healing (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 1 | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Recall phenomenon (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0
Blood gases abnormal (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0
General physical condition abnormal (Investigations) | 2 | 2 | 0 | 0
Influenza B virus test positive (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2 | 3 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 81 | 64 | 144 | 6
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 2 | 0 | 3 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 1 | 1
Cluster headache (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalitis autoimmune (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 2
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 0 | 0
Hemianopia homonymous (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Immune-mediated encephalitis (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 0 | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 1 | 0
Paresis (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 1 | 0
Transient aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 0 | 0
Device loosening (Product Issues) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 8 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast inflammation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 7 | 1
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 22 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 5 | 1
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 23 | 1 | 17 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 4 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 2 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eosinophilic cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Brachiocephalic vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2 | 2 | 0
Embolism (Vascular disorders) | 2 | 0 | 2 | 0
Exsanguination (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 3 | 0 | 1 | 0
Infarction (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 2 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=391) | Cohort A1 (N=198) | Cohort B (N=395) | Cohort C (N=57)
Anaemia (Blood and lymphatic system disorders) | 53 | 35 | 53 | 13
Atrial fibrillation (Cardiac disorders) | 13 | 6 | 8 | 3
Adrenal insufficiency (Endocrine disorders) | 9 | 4 | 7 | 4
Hyperthyroidism (Endocrine disorders) | 31 | 17 | 35 | 5
Hypothyroidism (Endocrine disorders) | 55 | 14 | 45 | 12
Dry eye (Eye disorders) | 7 | 1 | 4 | 4
Vision blurred (Eye disorders) | 10 | 6 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 33 | 5 | 21 | 7
Colitis (Gastrointestinal disorders) | 9 | 7 | 3 | 4
Constipation (Gastrointestinal disorders) | 69 | 26 | 53 | 11
Diarrhoea (Gastrointestinal disorders) | 122 | 48 | 80 | 23
Dry mouth (Gastrointestinal disorders) | 20 | 4 | 12 | 3
Dysphagia (Gastrointestinal disorders) | 12 | 4 | 11 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 1 | 3 | 4
Nausea (Gastrointestinal disorders) | 97 | 40 | 65 | 25
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 63 | 18 | 52 | 11
Asthenia (General disorders) | 84 | 45 | 67 | 4
Chills (General disorders) | 16 | 2 | 10 | 5
Fatigue (General disorders) | 140 | 39 | 87 | 24
Localised oedema (General disorders) | 0 | 1 | 0 | 4
Malaise (General disorders) | 7 | 1 | 3 | 3
Non-cardiac chest pain (General disorders) | 11 | 8 | 11 | 5
Oedema peripheral (General disorders) | 39 | 14 | 32 | 9
Pain (General disorders) | 20 | 6 | 10 | 5
Pyrexia (General disorders) | 66 | 25 | 51 | 7
Bronchitis (Infections and infestations) | 18 | 8 | 23 | 4
Nasopharyngitis (Infections and infestations) | 29 | 10 | 14 | 0
Pneumonia (Infections and infestations) | 23 | 15 | 17 | 4
Upper respiratory tract infection (Infections and infestations) | 23 | 6 | 23 | 6
Urinary tract infection (Infections and infestations) | 24 | 7 | 11 | 4
Fall (Injury, poisoning and procedural complications) | 12 | 2 | 8 | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 22 | 2 | 11 | 4
Alanine aminotransferase increased (Investigations) | 20 | 12 | 19 | 6
Amylase increased (Investigations) | 27 | 19 | 31 | 3
Aspartate aminotransferase increased (Investigations) | 14 | 11 | 18 | 6
Blood alkaline phosphatase increased (Investigations) | 10 | 8 | 20 | 6
Blood creatinine increased (Investigations) | 18 | 11 | 22 | 8
Lipase increased (Investigations) | 35 | 18 | 31 | 3
Lymphocyte count decreased (Investigations) | 3 | 0 | 2 | 3
Neutrophil count decreased (Investigations) | 3 | 1 | 4 | 3
Weight decreased (Investigations) | 33 | 16 | 23 | 8
Weight increased (Investigations) | 4 | 2 | 5 | 5
Decreased appetite (Metabolism and nutrition disorders) | 96 | 38 | 83 | 22
Dehydration (Metabolism and nutrition disorders) | 26 | 6 | 12 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 11 | 21 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 4 | 8 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 7 | 9 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 31 | 12 | 24 | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 4 | 4 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 18 | 13 | 29 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 | 25 | 44 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 7 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 51 | 15 | 47 | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 | 5 | 15 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 | 1 | 7 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 3 | 15 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 7 | 27 | 9
Dizziness (Nervous system disorders) | 32 | 15 | 24 | 7
Headache (Nervous system disorders) | 54 | 26 | 34 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 2 | 4
Anxiety (Psychiatric disorders) | 19 | 8 | 11 | 10
Depression (Psychiatric disorders) | 21 | 1 | 6 | 8
Insomnia (Psychiatric disorders) | 34 | 14 | 17 | 8
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 98 | 22 | 71 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 85 | 41 | 85 | 24
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 | 10 | 21 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 10 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 5 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 31 | 4 | 18 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 31 | 13 | 28 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 29 | 9 | 24 | 2
Erythema (Skin and subcutaneous tissue disorders) | 10 | 6 | 20 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 82 | 32 | 79 | 16
Rash (Skin and subcutaneous tissue disorders) | 59 | 31 | 52 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 30 | 6 | 16 | 10
Hypotension (Vascular disorders) | 20 | 5 | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT02869789/Prot_SAP_000.pdf